CLINICAL TRIAL: NCT05943548
Title: Omuyambi: Traditional Healer Support to Improve HIV Viral Suppression in Rural Uganda
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Mbarara University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-09025268; 1R01MH132440-01 (NIH)
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections
Keywords: Traditional Healer; Community Health
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: A parallel arm cluster randomized trial will be used to compare the effectiveness of the intervention to the control.
Masking Description: Masking is not possible due to the cluster randomized trial design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omuyambi Traditional Healer (TH) Intervention (Experimental): The traditional healer (TH) clusters randomized to the intervention arm will refer consented people living with HIV to a predetermined government-run HIV clinic for the provision of care. The patients that are in this arm will receive, adherence support for PLWH using a TH-tailored curriculum as an adjunct to clinic-based HIV care. These participants will also receive one-on-one counselling to improve self-efficacy, be provided social support, and will work with THs to develop individualized adherence strategies.
  Interventions: Behavioral: Omuyambi
- Control Arm (Placebo Comparator): The traditional healer (TH) clusters randomized to the control arm will refer consented people living with HIV to a predetermined government-run clinic for the provision of care. The patients in this arm will receive no additional linkage or psychosocial support.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Omuyambi — HIV testing, referral, care linkage, and medication adherence support
  Arms: Omuyambi Traditional Healer (TH) Intervention
Behavioral: Control — HIV Testing and referral
  Arms: Control Arm

SUMMARY:
This study aims to test a new approach to support people living with Human Immunodeficiency Virus (HIV) in Uganda. Traditional healers (TH) will be trained to provide counselling and testing for HIV, help patients start antiretroviral therapy quickly, and offer guidance on taking medications and staying in HIV care. This support will be given in addition to the regular care provided at clinics. The main goal of the study is to see if this new approach can help more people in rural areas achieve viral suppression.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old
* reactive point-of-care (POC) oral swab rapid HIV self-test (ex. OraQuick© HIV1/2 antibody testing) at the TH location or previously diagnosed with HIV (verified by the HIV clinic), and CASE adherence index score ≤10
* baseline viral load measurement of >200 copies/mL
* primary residence in Mbarara or Rwampara district
* agrees to study procedures, including that PLWH will go to one of the five pre-determined HIV clinics if they choose to receive HIV care, and in-person visits at baseline, 12- and 24-months with study nurse

Exclusion Criteria:

* Unwilling or unable to participate in study procedures or provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Viral Load Suppression in People Living with HIV (PLWH) at 12 months | 12 months
  Achievement and maintenance of HIV-1 RNA <200 copies/mL

SECONDARY OUTCOMES:
Linkage to HIV Care | 7 Days
  Number of PLWH linked to HIV care determined by completing one clinic visit within 7 days of study enrollment
Antiretroviral Therapy (ART) Initiation | 7 days
  Number of PLWH initiated on ART determined having (re)initiated ART within 7 days of study enrollment.
Antiretroviral Therapy (ART) Adherence | 12 months
  Number of PLWH adhering to ART determined by binary outcome of having dried blood spot (DBS) tenofovir diphosphate (TFV-DP) concentrations of ≥ 64 (adherence) or < 64 (non-adherence) nanograms per milliliter.
Retention in Care | 12 months
  Number of PLWH retaining care after 12 months. Defined as a binary outcome as attending the most recent appointment within 90 days of its scheduled date.
Medical Outcomes Study-HIV Health Survey (MOS-HIV) Score at 12 months | 12 months
  This scale evaluated perceived quality of life among people living with HIV. The scale is scored on a 0-100, with higher scores yielding better perceived quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Radhika Sundararajan, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and statistical analysis plan will be shared with any one who wishes to access the data beginning 3 months following and ending 5 years after article publication.
Supporting Information: Study Protocol, SAP
Time Frame: 3 months following and ending 5 years after article publication
Access Criteria: Researchers who propose a methodologically sound proposal to achieve aims in the approved proposal. Requesters will need to complete a data access agreement.

REFERENCES:
- [Derived] Hooda M, Stead M, Nuwagaba G, Natukunda S, Birungi C, Bugeza W, Tushabe M, Gogineni S, Nansera D, Muyindike W, Mwanga-Amumpaire J, Sundararajan R. 'Empowerment' as a proximal implementation outcome for task shifting with informal cadres: findings from a qualitative study with traditional healers in rural Uganda. Implement Sci Commun. 2025 Nov 29;7(1):3. doi: 10.1186/s43058-025-00823-9. PMID 41316446
- [Derived] Sundararajan R, Hooda M, Lai Y, Nansera D, Audet C, Downs J, Lee MH, McNairy M, Muyindike W, Mwanga-Amumpaire J. Traditional healer support to improve HIV viral suppression in rural Uganda (Omuyambi): study protocol for a cluster randomized hybrid effectiveness-implementation trial. Trials. 2024 Jul 1;25(1):430. doi: 10.1186/s13063-024-08286-4. PMID 38956628